CLINICAL TRIAL: NCT06672458
Title: Upper Extremity Functional Electrical Stimulation (FES) for Restoration of Upper Extremity Function After Spinal Cord Injury (SCI)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Matija Milosevic, Assistant Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20240966
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Spinal Cord Injuries; Peripheral Nerve Injuries
MeSH Terms: conditions — Spinal Cord Injuries; Peripheral Nerve Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Acute SCI Group (Experimental): Individuals with traumatic spinal cord injury (SCI) with a neurological level at or above T1 spinal cord level; Abbreviated Injury Scale (AIS) A, B, C or D impairment grade; less than 6 months post injury. Participants in this group will be in the study for up to 12 weeks
  Interventions: Device: MyndMove Short Term Therapy; Other: Conventional Short Term Therapy; Device: MyndMove Long Term Therapy
- Chronic SCI Group (Experimental): Individuals with traumatic spinal cord injury (SCI) with a neurological level at or above T1 spinal cord level; Abbreviated Injury Scale (AIS) A, B, C or D impairment grade; more than 6 months post injury. Participants in this group will be in the study for up to 12 weeks
  Interventions: Device: MyndMove Short Term Therapy; Other: Conventional Short Term Therapy; Device: MyndMove Long Term Therapy
- Acute PNI Group (Experimental): Individuals with PNI that are within 6 months pre- or post-UE nerve transfer surgery. Participants in this group will be in the study for up to 12 weeks
  Interventions: Device: MyndMove Short Term Therapy; Other: Conventional Short Term Therapy; Device: MyndMove Long Term Therapy
- Chronic PNI Group (Experimental): Individuals with PNI that are 6 months or more post-UE nerve transfer surgery. Participants in this group will be in the study for up to 12 weeks
  Interventions: Device: MyndMove Short Term Therapy; Other: Conventional Short Term Therapy; Device: MyndMove Long Term Therapy

INTERVENTIONS:
Device: MyndMove Short Term Therapy — FES therapy will be provided in one visit (one hour duration) delivered within a 2 week period, in person. FES therapy uses surface electrical stimulation to produce muscle contractions in different combinations to achieve a wide range of reaching and grasping functions. To achieve these movements the single use electrodes will be placed in various combinations on the surface of the different upper arm muscles. Participants will perform hand and finger dexterity tests as well as arm functional mobility tasks while receiving FES.
Other: Conventional Short Term Therapy — Therapy will be provided in one visit (one hour duration) delivered within a 2 week period, in person. Conventional therapy will consist of performance hand and finger dexterity tests as well as arm functional mobility tasks
Device: MyndMove Long Term Therapy — FES upper arm therapy will be provided in one-hour in-person sessions for a maximum of 40 sessions delivered no less than 3 times per week and up to 5 times per week during a period of up to 12 weeks. Over the course of 40 sessions, participants will progress through various movement sequences aimed at regaining natural, unassisted voluntary movements in the affected arms while receiving FES.

SUMMARY:
The purpose of this research is to examine the effects that functional electrical stimulation (FES) therapy has on the way the arms, brain and spinal cord work. The study team wants to understand what recovery looks like in persons with a spinal cord injury (SCI) or peripheral nerve injury (PNI) using the MyndMove (MyndTec Inc., Ontario, Canada) therapy system. This type of therapy uses stimulation to help people with SCI and other neurological conditions to perform common tasks, work out, or strengthen muscles.

ELIGIBILITY:
Inclusion Criteria:

1. Neurological Injury:

1. Traumatic spinal cord injury (SCI): neurological level at or above T1 spinal cord level; AIS A, B, C or D impairment grade

   * Group 1 (Acute SCI): Deemed medically stable by medical practitioner, less than 6 months post-injury.
   * Group 2 (Chronic SCI): More than 6 months post-injury.

   or
2. Peripheral nerve injury (PNI), with or without SCI, who are pre- or post- upper extremity (UE) nerve transfer surgery

   * Group 3 (Acute Pre- or Post-UE nerve transfer surgery): Deemed medically stable and safe/appropriate to participate in MyndMove UE FES therapy intervention by referring neurosurgeon within 6 months pre- or post-UE nerve transfer surgery.
   * Group 4 (Chronic Post-UE nerve transfer surgery): Deemed medically stable and safe/appropriate to participate in MyndMove UE FES therapy intervention by referring neurosurgeon 6 months or more post-UE nerve transfer surgery.

     3. Has detectable residual connection in upper-limb muscles in at least one of the neurologically affected sides confirmed by a visible contraction when functional electrical stimulation (FES) is applied in at least one upper extremity muscle at baseline.

     4. Has detectable motor function in at least 1 upper extremity muscle on 1 neurologically affected side confirmed by voluntary electromyography (EMG) or detectable motor evoked potential (MEP) at the baseline assessment. 5. (Aim 2 only) Able to commit to intervention and assessment sessions over a maximum duration of 4 months.

Exclusion Criteria

1. Traumatic brain injury, stroke, multiple sclerosis, or other disorders that could affect neuromotor function.
2. Severe spasticity that could prevent the study protocol as determined by the investigator.
3. Major executive dysfunction, dementia, depression, neurocognitive impairments, or other major medical co-morbidities.
4. Has contraindications for transcutaneous stimulation using FES such as breakdown of skin in the area that will come into contact with electrodes, thrombosis, or skin disease
5. Poorly managed autonomic dysreflexia that could be triggered by FES.
6. Unhealed upper extremity fracture, contracture, or pressure sore.
7. Implanted neurostimulator (e.g., deep brain stimulation (DBS), epidural/subdural, vagal nerve stimulation (VNS))
8. Cardiac pacemaker or intracardiac lines.
9. Individuals who require therapy or other care that could interfere with participation in the study.
10. Individuals on investigational drugs or any other intervention known to have a potential impact on neuromotor function.
11. Individuals with substance disorders, including alcoholism and drug abuse.
12. Individuals who are pregnant, breastfeeding, or the desire to become pregnant during the study.
13. In the opinion of the investigators, the study is not safe or appropriate for the participant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Nine Hole Peg Test | baseline and up to 2 weeks
  The Nine-Hole Peg Test assesses hand and finger dexterity. It is administered by asking the subject to take the pegs from a container, one by one, and place them into holes on the board as quickly as possible. Participants must then remove the pegs from the holes, one by one, and replace them back into the container. Test is performed at the beginning and end of each intervention visit. Scores are based on the time taken to complete the activity, recorded in seconds. (Only for subjects in short term intervention)
Surface EMG | baseline and up to 2 weeks
  EMG signals (measured in volts) recorded by skin surface EMG electrodes placed on the arm(s) during muscle contraction to evaluate muscle activity and motor unit activity at the beginning and end of each intervention visit. (Only for subjects in short term intervention)
Graded-Redefined Assessment of Strength, Sensibility, and Prehension (GRASSP) Prehension Performance (GR-PP) | baseline, 12 weeks
  GRASSP test will be used to assess upper arm motor function. Series of tasks will test subject's strength, sensation, and prehension. The prehension ability sub-test is scored for a total max score of 30 for each arm, using a scale from 0-30 where 0 is no upper arm motor function and 30 is full upper arm motor function. (Only for subjects in long term intervention)
Manual Muscle Test (MMT) with FES | baseline, 12 weeks
  A test that measures muscle strength and function with FES via MyndMove. Each muscle group tested (varies) will be scored from 0-5, where 0 is indicating no movement and strength and a max score of 5 indicating full, normal movement and strength. (Only for subjects in long term intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Matija Milosevic, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami - Miami Project to Cure Paralysis, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No